CLINICAL TRIAL: NCT02697734
Title: A Phase III, Multi-center, Randomized, Double-blind, 48 Week Study With an Initial 12 Week Placebo-controlled Period to Evaluate the Safety and Efficacy of Osilodrostat in Patients With Cushing's Disease
Brief Title: Efficacy and Safety Evaluation of Osilodrostat in Cushing's Disease
Acronym: LINC-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLCI699C2302
Record Dates: First submitted 2016-02-27; First posted 2016-03-03 (Estimated); Results first posted 2021-10-19 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Cushing's Disease
Keywords: Cushing's disease; LCI699; osilodrostat; Pituitary Gland; Adrenocorticotropic; Hormone; ACTH; UFC
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Pituitary Diseases | interventions — Osilodrostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- osilodrostat Group (Experimental): Participants in this arm were randomized to receive the study drug, osilodrostat followed after Week 12 by open-label osilodrostat at the starting dose (with a second dose titration)
  Interventions: Drug: osilodrostat
- osilodrostat Placebo Group (Placebo Comparator): Participants in this arm were randomized to receive osilodrostat placebo followed after Week 12 by open-label osilodrostat at the starting dose (with a dose titration)
  Interventions: Drug: osilodrostat Placebo

INTERVENTIONS:
Drug: osilodrostat — In the form of filmcoated tablets for oral administration, in the following dose strengths: 1 mg, 5 mg, 10 mg, and 20 mg.
  Other Names: LCI699
  Arms: osilodrostat Group
Drug: osilodrostat Placebo — Matching Placebo in the form of filmcoated tablets for oral administration
  Arms: osilodrostat Placebo Group

SUMMARY:
The purpose of this study was to confirm efficacy and safety of osilodrostat for the treatment of patients with Cushing's disease who are candidates for medical therapy.

DETAILED DESCRIPTION:
The study LCI699C2302 (LINC-4) is a multi-center, randomized, double-blind study to evaluate the safety and efficacy of osilodrostat in patients with Cushing's disease.

Enrolled patients were initially randomized to either osilodrostat or placebo, in a 2:1 ratio, for a 12-week double-blind period (Period 1). Randomization was stratified by history of pituitary radiation. After Week 12, all patients received open-label osilodrostat until the end of the Core phase at Week 48 (Period 2).

After Week 48, patients could join an optional 48 week extension period.

ELIGIBILITY:
Key inclusion criteria:

* Confirmed Cushing's Disease (CD) that is persistent or recurrent as evidenced by all of the following criteria being met (i.e., a, b and c):

  1. mUFC > 1.3 x ULN (Mean of three 24-hour urine samples collected preferably on 3 consecutive days, during screening after washout of prior medical therapy for CD (if applicable), confirmed by the central laboratory and available before Day 1), with ≥2 of the individual UFC values being > 1.3 x ULN.
  2. Morning plasma Adrenocorticotropic hormone (ACTH) above Lower Limit of Normal
  3. Confirmation (based on medical history) of pituitary source of excess

     ACTH as defined by any one or more of the following three criteria:

  i. Histopathologic confirmation of an ACTH-staining adenoma in patients who have had prior pituitary surgery. OR ii. Magnetic resonance imaging (MRI) confirmation of pituitary adenoma > 6 mm OR iii. Bilateral inferior petrosal sinus sampling (BIPSS) with either corticotropic-releasing hormone (CRH) or desmopressin (DDAVP) stimulation for patients with a tumor ≤ 6mm. The criteria for a confirmatory BIPSS test are any of the following: Pre-dose central to peripheral ACTH gradient > 2; Post-dose central to peripheral ACTH gradient > 3 after either CRH or DDAVP stimulation
* Patients that received glucocorticoid replacement therapy must have discontinued such therapy for at least seven days or 5 half-lives prior to screening, whichever is longer.
* Patients with de novo CD can be included only if they are not considered candidates for surgery (e.g., poor surgical candidates due to co-morbidities, inoperable tumors, patients who refuse to have surgical treatment, or surgical treatment is not available).

Key exclusion criteria:

* Patients with pseudo-Cushing's syndrome. This may be diagnosed by a normal late night salivary cortisol value collected during the screening period and after washout of prior CD medication.
* Patients with risk factors for QT corrected (QTc) prolongation or Torsade de Pointes, including:

patients with a baseline QT corrected (Fridericia QT formula) (QTcF) > 450 ms for males and QTcF > 460 ms for females; personal or family history of long QT syndrome; concomitant medications known to prolong the QT interval; patients with hypokalemia, hypocalcaemia, or hypomagnesaemia, if not corrected before pre-dose Day 1.

* Patients likely to require adrenalectomy, pituitary surgery, or radiation therapy during the placebo-controlled period (Weeks 1-12) for the treatment of severe hypercortisolism or pituitary tumor growth causing compression of the optic chiasm.
* Patients with compression of the optic chiasm due to a macroadenoma or patients at high risk of compression of the optic chiasm (tumor within 2 mm of optic chiasm).
* Patients who have a known inherited syndrome as the cause for hormone over secretion (i.e. Carney Complex, McCune-Albright syndrome, MEN-1, AIP).
* Patients with Cushing's syndrome due to ectopic ACTH secretion or ACTH independent (adrenal) Cushing's syndrome. Pregnant or nursing (lactating) women. 8. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 1 week after completion of dosing. Highly effective contraception methods include: A. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. B. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study drug. In case of bilateral oophorectomy, documentation is required (e.g. operative report, pelvic ultrasound or other reliable imaging method). C. Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.

D. Combination of any two of the following (a+b or a+c, or b+c):

1. Use of oral*, injected, or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository. *In the case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study drug. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child bearing potential.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (34):
- United States (6):
  - University of Colorado Endocrinology Clinical Trials Unit, Aurora, Colorado
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Columbia University Medical Center New York Presbyterian Neuroendocrine Unit, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health and Science University SC LCI699C2301, Portland, Oregon
  - University of Pennsylvania Medical Center University of Pennsylvania, Philadelphia, Pennsylvania
- Novartis Investigative Site, Leuven, Belgium
- Brazil (3):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- China (3):
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
- Novartis Investigative Site, San Pedro, San Jose, Costa Rica, Costa Rica
- Novartis Investigative Site, Athens, Greece
- Poland (3):
  - Novartis Investigative Site, Warsaw, Masovian Voivodeship
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, Porto, Portugal
- Novartis Investigative Site, Moscow, Russia
- Spain (6):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Lucerne, Switzerland
- Thailand (2):
  - Novartis Investigative Site, Bangkok, THA
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Fleseriu M, Pivonello R, Lacroix A, Biller BMK, Feelders R, Gadelha M, Bertherat J, Belaya Z, Piacentini A, Pedroncelli AM, Newell-Price J. Osilodrostat dose impact on efficacy/safety in Cushing's disease: large, pooled analysis of LINC 2, 3, and 4. Eur J Endocrinol. 2025 Oct 30;193(5):606-617. doi: 10.1093/ejendo/lvaf207. PMID 41052284
- [Derived] Newell-Price J, Fleseriu M, Pivonello R, Feelders RA, Gadelha MR, Lacroix A, Witek P, Heaney AP, Piacentini A, Pedroncelli AM, Biller BMK. Improved Clinical Outcomes During Long-term Osilodrostat Treatment of Cushing Disease With Normalization of Late-night Salivary Cortisol and Urinary Free Cortisol. J Endocr Soc. 2024 Nov 12;9(1):bvae201. doi: 10.1210/jendso/bvae201. eCollection 2024 Nov 26. PMID 39610378
- [Derived] Gadelha M, Bex M, Feelders RA, Heaney AP, Auchus RJ, Gilis-Januszewska A, Witek P, Belaya Z, Yu Y, Liao Z, Ku CHC, Carvalho D, Roughton M, Wojna J, Pedroncelli AM, Snyder PJ. Randomized Trial of Osilodrostat for the Treatment of Cushing Disease. J Clin Endocrinol Metab. 2022 Jun 16;107(7):e2882-e2895. doi: 10.1210/clinem/dgac178. PMID 35325149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set: comprises all randomized participants who received at least one dose of study drug (osilodrostat or placebo).
  There are 73 participants in the FAS who were randomized and received treatment.
Groups:
- Osilodrostat Group: Participants in this arm were randomized to receive the study drug, osilodrostat, followed after Week 12 by open-label osilodrostat at the starting dose (with a second dose titration).
Period: Core Phase - up to Week 48
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Started (treated) | 48 | 25
Completed | 42 | 23
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 1 | 0
Period: Optional Extension Phase
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Started | 38 | 22
Completed | 33 | 20
Not Completed | 5 | 2
Not completed — Adverse Event | 5 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group | Total
Number analyzed (Participants) | 48 | 25 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 25 | 71
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Participants
  Years | 42.3 (13.82) | 38.9 (12.33) | 41.2 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 18 | 61
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 34 | 15 | 49
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Randomized Participants With a Complete Response
Description: A complete responder at week 12 is defined as a participant who had a mean urine free cortisol ≤ upper limit of normal (mUFC ≤ ULN) at Week 12.
  Participants who had a missing mUFC assessment at Week 12 were counted as non-responders for the primary endpoint.
Time Frame: at Week 12
Population: Full Analysis Set: comprises all randomized participants who received at least one dose of study drug (osilodrostat or placebo)
Measure: Count of Participants; unit: Participants
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
Participants | 37 | 2
Statistical Analysis 1: Comparison: Osilodrostat Group vs Osilodrostat Placebo Group; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 43.4, 95% CI 2-sided [7.06 to 343.19]

2. Secondary Outcome: Percentage of Participants With mUFC ≤ ULN at Week 36
Description: The complete response rate in both arms combined at Week 36. A complete responder at Week 36 is defined as a participant who had mean urine free cortisol <= upper limit of normal (mUFC <= ULN) at Week 36. Participants with missing mUFC at Week 36 were counted as non-responders.
Time Frame: At Week 36
Population: Full Analysis Set participants: comprises all randomized participants who received at least one dose of osilodrostat. Only a single arm is reported since the endpoint is 'To assess the complete response rate in both arms combined at Week 36 in patients receiving osilodrostat treatment.'
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Participants Combined: Consisted of all randomized participants who received at least one dose of osilodrostat.
Arm/Group | All Participants Combined
Number analyzed (Participants) | 73
Percentage of participants | 80.8 [69.9 to 89.1]

3. Secondary Outcome: Change From Baseline in mUFC
Description: To assess the change in mean urinary free cortisol (mUFC) from baseline by treatment arm.
Time Frame: Baseline, weeks 2,5,8,12,14,17,20,23,26,29,32,36,40,48,60,72,84,96
Population: Full Analysis Set: comprises all randomized participants who received at least one dose of study drug (osilodrostat or placebo). The number analyzed varied from one visit to another because of missed visits, missed assessments, early discontinuation from the study, and completion of the extension phase.
Measure: Mean (Standard Deviation); unit: nmol/24hr
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
nmol/24hr
  actual - baseline | 421.4 (291.25) | 451.5 (535.09)
  change from baseline at week 2 (n=47,24): number analyzed (Participants) | 47 | 24
  change from baseline at week 2 (n=47,24) | -139.3 (404.45) | 164.9 (543.82)
  change from baseline at week 5 (n=46,25): number analyzed (Participants) | 46 | 25
  change from baseline at week 5 (n=46,25) | -252.8 (338.48) | -37.3 (280.84)
  change from baseline at week 8 (n=44,25): number analyzed (Participants) | 44 | 25
  change from baseline at week 8 (n=44,25) | -330.2 (303.35) | -35.0 (325.30)
  change from baseline at week 12 (n=44,24): number analyzed (Participants) | 44 | 24
  change from baseline at week 12 (n=44,24) | -332.7 (315.50) | -49.1 (332.29)
  change from baseline at week 14 (n=45,25): number analyzed (Participants) | 45 | 25
  change from baseline at week 14 (n=45,25) | -191.7 (446.77) | -209.5 (407.62)
  change from baseline at week 17 (n=45,25): number analyzed (Participants) | 45 | 25
  change from baseline at week 17 (n=45,25) | -238.8 (362.46) | -284.5 (557.47)
  change from baseline at week 20 (n=44,24): number analyzed (Participants) | 44 | 24
  change from baseline at week 20 (n=44,24) | -294.5 (316.65) | -355.1 (538.96)
  change from baseline at week 23 (n=44,25): number analyzed (Participants) | 44 | 25
  change from baseline at week 23 (n=44,25) | -314.1 (307.60) | -387.8 (466.15)
  change from baseline at week 26 (n=43,25): number analyzed (Participants) | 43 | 25
  change from baseline at week 26 (n=43,25) | -345.2 (306.35) | -365.4 (458.28)
  change from baseline at week 29 (n=43,25): number analyzed (Participants) | 43 | 25
  change from baseline at week 29 (n=43,25) | -331.4 (299.63) | -391.4 (534.57)
  change from baseline at week 32 (n=44,25): number analyzed (Participants) | 44 | 25
  change from baseline at week 32 (n=44,25) | -341.3 (298.96) | -298.0 (655.52)
  change from baseline at week 36 (n=43,25): number analyzed (Participants) | 43 | 25
  change from baseline at week 36 (n=43,25) | -349.6 (310.46) | -372.9 (519.17)
  change from baseline at week 40 (n=43,23): number analyzed (Participants) | 43 | 23
  change from baseline at week 40 (n=43,23) | -333.4 (307.63) | -364.7 (542.28)
  change from baseline at week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  change from baseline at week 48 (n=42,22) | -325.1 (314.30) | -367.5 (554.16)
  change from baseline at week 60 (n=33,19): number analyzed (Participants) | 33 | 19
  change from baseline at week 60 (n=33,19) | -364.4 (339.57) | -335.2 (571.06)
  change from baseline at week 72 (n=31,17): number analyzed (Participants) | 31 | 17
  change from baseline at week 72 (n=31,17) | -381.2 (338.68) | -372.4 (624.69)
  change from baseline at week 84 (n=23,17): number analyzed (Participants) | 23 | 17
  change from baseline at week 84 (n=23,17) | -398.6 (377.81) | -196.0 (916.83)
  change from baseline at week 96 (n=6,7): number analyzed (Participants) | 6 | 7
  change from baseline at week 96 (n=6,7) | -414.5 (347.83) | -616.4 (881.92)

4. Secondary Outcome: Time-to-first Control of mUFC - Number (%) of Participants With mUFC <=ULN
Description: To assess time-to-first control of mUFC, (in days) from randomization to the first mUFC collection that was ≤ ULN before completion/discontinuation of placebo-controlled period.
  Participants who did not achieve post-baseline mUFC control were censored at discontinuation or completion of placebo-controlled period, whichever was earlier.
Time Frame: up to 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
Participants | 45 | 8

5. Secondary Outcome: Time-to-first Control of mUFC - Median Time to First Controlled mUFC Response
Description: To assess time-to-first control of mUFC, (in days) from randomization to the first mUFC collection that was ≤ ULN before completion/discontinuation of placebo-controlled period.
  Participants who did not achieve post-baseline mUFC control were censored at discontinuation or completion of placebo-controlled period, whichever was earlier.
  The median time-to-first control and corresponding two-sided 95% Confidence Interval were calculated using Kaplan-Meier methodology of Brookmeyer and Crowley (1982).
Time Frame: up to 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
Days | 35 [34.0 to 52.0] | NA [87.0 to NA] — Not estimable. Due to the low number of participants achieving control in the placebo arm, median time-to-first control was not reached and the median with corresponding upper 95% confidence interval could not be estimated.

6. Secondary Outcome: Time-to-first Control of mUFC - % Event Probability Estimates
Description: To assess time-to-first control of mUFC, (in days) from randomization to the first mUFC collection that was ≤ ULN before completion/discontinuation of placebo-controlled period.
  Participants who did not achieve post-baseline mUFC control were censored at discontinuation or completion of placebo-controlled period, whichever was earlier.
  % Event probability estimate is the estimated probability that a participant will have an event prior to the specified time point. % Event probability estimates are obtained from the Kaplan-Meier survival estimates for all treatment groups; Greenwood formula is used for Confidence Interval (CI) of Kaplan-Meier (KM) estimates.
Time Frame: up to 12 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent (event probability estimates)
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
Percent (event probability estimates)
  2 Weeks | 25.0 [15.0 to 39.8] | 16.0 [6.3 to 37.2]
  5 Weeks | 60.4 [47.0 to 74.1] | 20.0 [8.9 to 41.6]
  8 Weeks | 79.4 [67.0 to 89.4] | 28.0 [14.5 to 49.9]
  12 Weeks | NA [NA to NA] — Not estimable as not reached | 28.0 [14.5 to 49.9]

7. Secondary Outcome: Time-to-escape During Osilodrostat Treatment From Collection of Normal mUFC (≤ ULN) to the First mUFC > 1.3 x ULN - Number (%) of Participants
Description: To assess time-to-escape from the first collection of normal mUFC (≤ ULN) to the first mUFC > 1.3 x ULN on two consecutive visits on the highest tolerated dose of osilodrostat and not related to a dose interruption or dose reduction due to safety reasons. Escape will not be assessed for participants during the first 26 weeks.
Time Frame: up to 48 weeks
Population: Full Analysis Set: comprises all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All Participants
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group | All Participants
Number analyzed (Participants) | 48 | 25 | 73
Participants | 0 | 2 | 2

8. Secondary Outcome: Time-to-escape During Osilodrostat Treatment From Collection of Normal mUFC (≤ ULN) to the First mUFC > 1.3 x ULN - Median Time to Escape From Normal mUFC
Description: To assess time-to-escape from the first collection of normal mUFC (≤ ULN) to the first mUFC > 1.3 x ULN on two consecutive visits on the highest tolerated dose of osilodrostat and not related to a dose interruption or dose reduction due to safety reasons. Escape will not be assessed for participants during the first 26 weeks.
  The median time-to-escape and corresponding two-sided 95% Confidence Interval were calculated using Kaplan-Meier methodology of Brookmeyer and Crowley (1982).
Time Frame: from week 26 to week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group | All Participants
Number analyzed (Participants) | 48 | 25 | 73
days | NA [NA to NA] — Not estimable as not reached due to the low number of events. | NA [116.0 to NA] — Not estimable as not reached due to the low number of events. | NA [NA to NA] — Not estimable as not reached due to the low number of events.

9. Secondary Outcome: Time-to-escape During Osilodrostat Treatment From Collection of Normal mUFC (≤ ULN) to the First mUFC > 1.3 x ULN - % Event Probability Estimates
Description: Escape is defined as the first loss of control of urinary free cortisol (UFC) that meets all of the following criteria: 1. prior normalization of UFC has occurred (median urinary free cortisol (mUFC)≤ upper limit of normal (ULN)); 2. patient reached the highest tolerated dose of osilodrostat; 3. 2 consecutive mUFC (collected at scheduled visits) were above 1.3x ULN; 4. the loss of control of UFC is not related to a dose interruption or dose reduction due to safety reasons; 5. happened beyond Week 26 when the patients have a chance to be treated with doses as high as 30 mg bid.
  * Event probability estimate is the estimated probability that a participant will have an event prior to the specified time point.
  * Event probability estimates are obtained from the Kaplan-Meier survival estimates for all treatment groups; Greenwood formula is used for CI of KM estimates.
Time Frame: week 26 and week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent (event probability estimates)
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group | All Participants
Number analyzed (Participants) | 48 | 25 | 73
Percent (event probability estimates)
  % Event probability estimates (95% CI) at 26 Weeks | 0 [NA to NA] — Not estimable as not reached due to the low number of events | 21.3 [5.7 to 61.9] | 15.6 [4.1 to 49.6]
  % Event probability estimates (95% CI) at 36 Weeks | 0 [NA to NA] — Not estimable as not reached due to the low number of events | NA [NA to NA] — Not estimable as not reached due to the low number of events | 15.6 [4.1 to 49.6]

10. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) by Dual-energy X-ray Absorptiometry (DXA) Scan at the Femoral Neck, Hip and Spinal Cord - QC Corrected
Description: The change from baseline in bone mineral density at the femoral neck, hip and spinal cord at Week 48 by treatment arm - QC corrected. An increase in bone mineral density is indicative of an improvement.
Time Frame: Baseline, week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 43 | 24
g/cm2
  FEMORAL NECK QC CORRECTED - baseline - Actual (n=43,24) | 0.8 (0.16) | 0.8 (0.14)
  FEMORAL NECK QC CORRECTED - week 48 - Actual change from baseline (n=28,19): number analyzed (Participants) | 28 | 19
  FEMORAL NECK QC CORRECTED - week 48 - Actual change from baseline (n=28,19) | 0.0 (0.04) | 0.0 (0.03)
  HIP QC CORRECTED - baseline - Actual (n=43,24) | 0.9 (0.14) | 0.9 (0.11)
  HIP QC CORRECTED - week 48 - Actual change from baseline (n=28,19): number analyzed (Participants) | 28 | 19
  HIP QC CORRECTED - week 48 - Actual change from baseline (n=28,19) | 0.0 (0.03) | 0.0 (0.02)
  SPINAL CORD QC CORRECTED - baseline - Actual (n=42,23): number analyzed (Participants) | 42 | 23
  SPINAL CORD QC CORRECTED - baseline - Actual (n=42,23) | 1.0 (0.15) | 1.0 (0.18)
  SPINAL CORD QC CORRECTED - week 48 - Actual change from baseline (n=28,18): number analyzed (Participants) | 28 | 18
  SPINAL CORD QC CORRECTED - week 48 - Actual change from baseline (n=28,18) | 0.0 (0.04) | 0.0 (0.04)

11. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) T-score by Dual-energy X-ray Absorptiometry (DXA) Scan at the Femoral Neck, Hip and Spinal Cord - QC Corrected
Description: The change from baseline in bone mineral density at the femoral neck, hip and spinal cord at Week 48 by treatment arm - QC corrected. An increase in bone mineral density is indicative of an improvement. T-score is the number of standard deviations above or below the mean for a healthy 30-year-old adult of the same sex and ethnicity as the patient. The WHO criteria are: Normal is a T-score of -1.0 or higher"
Time Frame: Baseline, week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 43 | 24
scores on a scale
  FEMORAL NECK QC CORRECTED - baseline - Actual (n=43,24) | -1.2 (1.06) | -1.3 (0.89)
  FEMORAL NECK QC CORRECTED - Actual change from baseline at week 48 (n=28,19): number analyzed (Participants) | 28 | 19
  FEMORAL NECK QC CORRECTED - Actual change from baseline at week 48 (n=28,19) | 0.1 (0.30) | 0.1 (0.21)
  HIP QC CORRECTED - baseline - Actual (n=43,24) | -0.7 (1.08) | -0.8 (0.84)
  HIP QC CORRECTED - Actual change from baseline at week 48 (n=28,19): number analyzed (Participants) | 28 | 19
  HIP QC CORRECTED - Actual change from baseline at week 48 (n=28,19) | 0.0 (0.27) | 0.0 (0.16)
  SPINAL CORD QC CORRECTED - baseline - Actual (n=42,23): number analyzed (Participants) | 42 | 23
  SPINAL CORD QC CORRECTED - baseline - Actual (n=42,23) | -1.2 (1.10) | -1.1 (1.40)
  SPINAL CORD QC CORRECTED - Actual change from baseline at week 48 (n=28,18): number analyzed (Participants) | 28 | 18
  SPINAL CORD QC CORRECTED - Actual change from baseline at week 48 (n=28,18) | 0.1 (0.32) | 0.1 (0.33)

12. Secondary Outcome: Patients With a Complete Response (mUFC ≤ ULN) or a Partial Response (mUFC Decrease ≥ 50% From Baseline and >ULN) at Week 12, 36 and 48
Description: Overall response rate defined as percentage of complete responders (mUFC ≤ ULN) plus partial responders (≥ 50% reduction in mUFC from baseline and >ULN) at week 12, 36, 48 by treatment arms for all patients.
Time Frame: baseline, week 12, 36 and 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
Participants
  week 12 Complete responders | 37 | 2
  week 12 Partial responders | 2 | 2
  week 12 Overall responders (complete or partial responders) | 39 | 4
  week 12 Non-responders | 9 | 21
  week 36 Complete responders | 38 | 21
  week 36 Partial responders | 2 | 3
  week 36 Overall responders (complete or partial responders) | 40 | 24
  week 36 Non-responders | 8 | 1
  week 48 Complete responders | 34 | 16
  week 48 Partial responders | 5 | 3
  week 48 Overall responders (complete or partial responders) | 39 | 19
  week 48 Non-responders | 9 | 6

13. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change from baseline in fasting plasma glucose at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 47 | 24
mg/dL
  Fasting glucose (mg/dL) - baseline - actual (n=47,24) | 97.3 (18.14) | 91.4 (15.15)
  Fasting glucose (mg/dL) - change from baseline at week 12 (n=44,23): number analyzed (Participants) | 44 | 23
  Fasting glucose (mg/dL) - change from baseline at week 12 (n=44,23) | -4.3 (14.84) | -1.7 (10.59)
  Fasting glucose (mg/dL) - change from baseline at week 36 (n=43,24): number analyzed (Participants) | 43 | 24
  Fasting glucose (mg/dL) - change from baseline at week 36 (n=43,24) | -6.7 (12.48) | -1.1 (12.93)
  Fasting glucose (mg/dL) - change from baseline at week 48 (n=41,21): number analyzed (Participants) | 41 | 21
  Fasting glucose (mg/dL) - change from baseline at week 48 (n=41,21) | -5.6 (14.13) | 1.8 (13.92)

14. Secondary Outcome: Change in Hemoglobin A1C
Description: Change from baseline in Hemoglobin A1C (%) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of Hemoglobin A1C
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
percentage of Hemoglobin A1C
  Hemoglobin A1C (%) - Actual - baseline | 6.0 (0.92) | 5.7 (0.56)
  Hemoglobin A1C (%) - Actual change from baseline at week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Hemoglobin A1C (%) - Actual change from baseline at week 12 (n=46,24) | -0.2 (0.44) | 0.0 (0.27)
  Hemoglobin A1C (%) Actual change from baseline at week 36 (n=44,25): number analyzed (Participants) | 44 | 25
  Hemoglobin A1C (%) Actual change from baseline at week 36 (n=44,25) | -0.2 (0.54) | -0.1 (0.46)
  Hemoglobin A1C (%) Actual change from baseline at week 48 (n=41,21): number analyzed (Participants) | 41 | 21
  Hemoglobin A1C (%) Actual change from baseline at week 48 (n=41,21) | -0.2 (0.58) | 0.1 (0.37)

15. Secondary Outcome: Change in Cholesterol
Description: Change from baseline in Cholesterol (mmol/L) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 45 | 25
mmol/L
  Cholesterol (mmol/L) - actual - baseline (n=45,25) | 5.7 (1.30) | 5.3 (1.15)
  Cholesterol (mmol/L) - change from baseline at week 12 (n=44,24): number analyzed (Participants) | 44 | 24
  Cholesterol (mmol/L) - change from baseline at week 12 (n=44,24) | -0.8 (0.95) | 0.0 (0.65)
  Cholesterol (mmol/L) - change from baseline at week 36 (n=44,25): number analyzed (Participants) | 44 | 25
  Cholesterol (mmol/L) - change from baseline at week 36 (n=44,25) | -1.0 (1.28) | -0.4 (0.89)
  Cholesterol (mmol/L) - change from baseline at week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Cholesterol (mmol/L) - change from baseline at week 48 (n=42,22) | -0.6 (1.36) | -0.4 (1.18)

16. Secondary Outcome: Change in LDL Cholesterol
Description: Change from baseline in LDL Cholesterol (mmol/L) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 45 | 24
mmol/L
  LDL Cholesterol (mmol/L) - Actual - baseline (n=45,24) | 3.4 (1.12) | 3.0 (1.07)
  LDL Cholesterol (mmol/L) - Actual change from baseline at week 12 (n=44,23): number analyzed (Participants) | 44 | 23
  LDL Cholesterol (mmol/L) - Actual change from baseline at week 12 (n=44,23) | -0.5 (0.80) | 0.1 (0.47)
  LDL Cholesterol (mmol/L) - Actual change from baseline at week 36 (n=44,24): number analyzed (Participants) | 44 | 24
  LDL Cholesterol (mmol/L) - Actual change from baseline at week 36 (n=44,24) | -0.6 (1.08) | -0.2 (0.70)
  LDL Cholesterol (mmol/L) - Actual change from baseline at week 48 (n=41,21): number analyzed (Participants) | 41 | 21
  LDL Cholesterol (mmol/L) - Actual change from baseline at week 48 (n=41,21) | -0.5 (0.99) | -0.2 (0.92)

17. Secondary Outcome: Change in HDL Cholesterol
Description: Change from baseline in HDL Cholesterol (mmol/L) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 45 | 25
mmol/L
  HDL Cholesterol (mmol/L) - Actual - baseline (n=45,25) | 1.6 (0.35) | 1.5 (0.38)
  HDL Cholesterol (mmol/L) - Actual change from baseline at week 12 (n=44,24): number analyzed (Participants) | 44 | 24
  HDL Cholesterol (mmol/L) - Actual change from baseline at week 12 (n=44,24) | -0.3 (0.29) | 0.0 (0.28)
  HDL Cholesterol (mmol/L) - Actual change from baseline at week 36 (n=44,25): number analyzed (Participants) | 44 | 25
  HDL Cholesterol (mmol/L) - Actual change from baseline at week 36 (n=44,25) | -0.3 (0.27) | -0.2 (0.25)
  HDL Cholesterol (mmol/L) - Actual - change from baseline at week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  HDL Cholesterol (mmol/L) - Actual - change from baseline at week 48 (n=42,22) | -0.2 (0.27) | -0.1 (0.29)

18. Secondary Outcome: Change in Triglyceride
Description: Change from baseline in Triglyceride (mmol/L) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 45 | 25
mmol/L
  Triglyceride (mmol/L) - Actual - baseline (n=45,25) | 1.5 (0.79) | 1.7 (0.85)
  Triglyceride (mmol/L) - Actual change from baseline at week 12(n=44,24): number analyzed (Participants) | 44 | 24
  Triglyceride (mmol/L) - Actual change from baseline at week 12(n=44,24) | 0.0 (0.53) | -0.2 (0.54)
  Triglyceride (mmol/L) - Actual change from baseline at week 36 (n=44,25): number analyzed (Participants) | 44 | 25
  Triglyceride (mmol/L) - Actual change from baseline at week 36 (n=44,25) | -0.1 (0.55) | -0.1 (0.71)
  Triglyceride (mmol/L) - Actual change from baseline at week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Triglyceride (mmol/L) - Actual change from baseline at week 48 (n=42,22) | 0.1 (0.92) | -0.2 (0.62)

19. Secondary Outcome: Change in Standing Systolic Blood Pressure
Description: Change from baseline in Standing Systolic Blood Pressure (mmHg) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 46 | 25
mmHg
  Standing Systolic Blood Pressure (mmHg) - Actual - baseline (n=46,25) | 132.4 (19.16) | 130.0 (17.72)
  Standing Systolic Blood Pressure (mmHg) - Actual change from baseline at week 12 (n=44,24): number analyzed (Participants) | 44 | 24
  Standing Systolic Blood Pressure (mmHg) - Actual change from baseline at week 12 (n=44,24) | -7.1 (18.08) | -0.9 (11.77)
  Standing Systolic Blood Pressure (mmHg) - Actual change from baseline at week 36 (n=42,25): number analyzed (Participants) | 42 | 25
  Standing Systolic Blood Pressure (mmHg) - Actual change from baseline at week 36 (n=42,25) | -9.3 (19.09) | -7.0 (21.04)
  Standing Systolic Blood Pressure (mmHg) - Actual change from baseline at week 48 (n=41,22): number analyzed (Participants) | 41 | 22
  Standing Systolic Blood Pressure (mmHg) - Actual change from baseline at week 48 (n=41,22) | -9.1 (19.45) | -11.0 (22.30)

20. Secondary Outcome: Change in Supine Systolic Blood Pressure
Description: Change from baseline in Supine Systolic Blood Pressure (mmHg) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
mmHg
  Supine Systolic Blood Pressure (mmHg) - Actual - baseline (n=48,25) | 131.7 (18.33) | 127.8 (18.69)
  Supine Systolic Blood Pressure (mmHg) - Actual change from baseline at week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Supine Systolic Blood Pressure (mmHg) - Actual change from baseline at week 12 (n=46,24) | -8.0 (17.54) | 2.3 (15.91)
  Supine Systolic Blood Pressure (mmHg) - Actual change from baseline at week 36 (n=42,25): number analyzed (Participants) | 42 | 25
  Supine Systolic Blood Pressure (mmHg) - Actual change from baseline at week 36 (n=42,25) | -9.7 (19.88) | -4.4 (17.43)
  Supine Systolic Blood Pressure (mmHg) - Actual change from baseline at week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Supine Systolic Blood Pressure (mmHg) - Actual change from baseline at week 48 (n=42,22) | -7.4 (19.38) | -7.5 (18.91)

21. Secondary Outcome: Change in Standing Diastolic Blood Pressure
Description: Change from baseline in Standing Diastolic Blood Pressure (mmHg) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 46 | 25
mmHg
  Standing Diastolic Blood Pressure (mmHg) - Actual - baseline (n=46,25) | 87.2 (12.74) | 88.2 (10.83)
  Standing Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 12 (n=44,24): number analyzed (Participants) | 44 | 24
  Standing Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 12 (n=44,24) | -4.8 (11.14) | -1.4 (9.84)
  Standing Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 36 (n=42,25): number analyzed (Participants) | 42 | 25
  Standing Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 36 (n=42,25) | -6.0 (12.09) | -4.4 (13.98)
  Standing Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 48 (n=41,22): number analyzed (Participants) | 41 | 22
  Standing Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 48 (n=41,22) | -4.4 (11.64) | -3.9 (13.36)

22. Secondary Outcome: Change in Supine Diastolic Blood Pressure
Description: Change from baseline in Supine Diastolic Blood Pressure (mmHg) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
mmHg
  Supine Diastolic Blood Pressure (mmHg) - Actual - baseline (n=48,25) | 83.9 (11.71) | 81.4 (11.21)
  Supine Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Supine Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 12 (n=46,24) | -6.3 (11.05) | -0.1 (8.31)
  Supine Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 36 (n=44,25): number analyzed (Participants) | 44 | 25
  Supine Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 36 (n=44,25) | -7.7 (11.92) | -3.4 (11.37)
  Supine Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 48 (n=41,22): number analyzed (Participants) | 41 | 22
  Supine Diastolic Blood Pressure (mmHg) - Actual change from baseline at week 48 (n=41,22) | -5.8 (11.60) | -3.7 (10.92)

23. Secondary Outcome: Change in Weight
Description: Change from baseline in Weight (kg) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
kg
  Weight (kg) - Actual - baseline (n=48,25) | 78.8 (17.46) | 77.3 (16.90)
  Weight (kg) - Actual change from baseline at week 12(n=46,24): number analyzed (Participants) | 46 | 24
  Weight (kg) - Actual change from baseline at week 12(n=46,24) | -0.8 (3.09) | -0.1 (2.12)
  Weight (kg) - Actual change from baseline at week 36 (n=44,25): number analyzed (Participants) | 44 | 25
  Weight (kg) - Actual change from baseline at week 36 (n=44,25) | -3.0 (5.53) | -4.8 (5.63)
  Weight (kg) - Actual change from baseline at week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Weight (kg) - Actual change from baseline at week 48 (n=42,22) | -3.6 (6.53) | -5.5 (6.38)

24. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline in Waist Circumference (cm) at Week 12, Week 36, and Week 48 by treatment arm
Time Frame: Baseline, weeks 12, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
cm
  Waist Circumference (cm)) - Actual - baseline (n=48,25) | 102.5 (17.01) | 103.4 (15.52)
  Waist Circumference (cm) - Actual change from baseline at week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Waist Circumference (cm) - Actual change from baseline at week 12 (n=46,24) | -1.0 (4.43) | -0.5 (3.35)
  Waist Circumference (cm)) - Actual change from baseline at week 36 (n=44,25): number analyzed (Participants) | 44 | 25
  Waist Circumference (cm)) - Actual change from baseline at week 36 (n=44,25) | -3.9 (6.36) | -2.1 (8.60)
  Waist Circumference (cm) - Actual change from baseline at week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Waist Circumference (cm) - Actual change from baseline at week 48 (n=42,22) | -4.1 (6.10) | -5.3 (5.68)

25. Secondary Outcome: Change From Baseline to Week 12, Week 36, and Week 48 in Clinical Signs of Cushing's Disease
Description: Change from baseline to Week 12, Week 36, and Week 48 in each of the following clinical signs of Cushing's disease, captured by: a semi-quantitative Likert scale for facial rubor, striae, supraclavicular fat pad, dorsal fat pad, proximal muscle wasting (atrophy), central (abdominal) obesity, and ecchymoses (bruises) by randomized treatment arm. The number/proportion of participants with an improvement or no change compared to baseline are reported
Time Frame: baseline, Week 12, Week 36 and Week 48
Population: Full Analysis Set: comprises all randomized participants who received at least one dose of study drug (osilodrostat or placebo). The number analyzed varied from one visit to another because of missed visits, missed assessments, early discontinuation from the study, and completion of the extension phase. Values for improvement or no change are reported. Hirsutism applies only to females, and thus the number analyzed is lower than for other clinical signs.
Measure: Count of Participants; unit: Participants
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 42 | 24
Participants
  Facial Rubor - week 12 (n=42,20): number analyzed (Participants) | 42 | 20
  Facial Rubor - week 12 (n=42,20) | 36 | 19
  Hirsutism - week 12 (n=36,16): number analyzed (Participants) | 36 | 16
  Hirsutism - week 12 (n=36,16) | 34 | 15
  Striae - week 12 (n=41,20): number analyzed (Participants) | 41 | 20
  Striae - week 12 (n=41,20) | 38 | 19
  Supraclavicular Fat Pad - week 12 (n=42,21): number analyzed (Participants) | 42 | 21
  Supraclavicular Fat Pad - week 12 (n=42,21) | 41 | 19
  Dorsal Fat Pad - week 12 (n=41,21): number analyzed (Participants) | 41 | 21
  Dorsal Fat Pad - week 12 (n=41,21) | 35 | 17
  Proximal Muscle Atrophy - week 12 (n=42,21): number analyzed (Participants) | 42 | 21
  Proximal Muscle Atrophy - week 12 (n=42,21) | 38 | 20
  Central Obesity - week 12 (n=42,21): number analyzed (Participants) | 42 | 21
  Central Obesity - week 12 (n=42,21) | 37 | 21
  Ecchymoses - week 12 (n=42,20): number analyzed (Participants) | 42 | 20
  Ecchymoses - week 12 (n=42,20) | 39 | 19
  Facial Rubor - week 36 (n=41,23): number analyzed (Participants) | 41 | 23
  Facial Rubor - week 36 (n=41,23) | 39 | 22
  Hirsutism - week 36 (n=34,17): number analyzed (Participants) | 34 | 17
  Hirsutism - week 36 (n=34,17) | 28 | 16
  Striae - week 36 (n=40,23): number analyzed (Participants) | 40 | 23
  Striae - week 36 (n=40,23) | 38 | 23
  Supraclavicular Fat Pad - week 36 (n=41,24): number analyzed (Participants) | 41 | 24
  Supraclavicular Fat Pad - week 36 (n=41,24) | 40 | 24
  Dorsal Fat Pad - week 36 (n=40,24): number analyzed (Participants) | 40 | 24
  Dorsal Fat Pad - week 36 (n=40,24) | 36 | 22
  Proximal Muscle Atrophy - week 36 (n=41,23): number analyzed (Participants) | 41 | 23
  Proximal Muscle Atrophy - week 36 (n=41,23) | 37 | 22
  Central Obesity - week 36 (n=41,24): number analyzed (Participants) | 41 | 24
  Central Obesity - week 36 (n=41,24) | 37 | 21
  Ecchymoses - week 36 (n=41,23): number analyzed (Participants) | 41 | 23
  Ecchymoses - week 36 (n=41,23) | 39 | 22
  Facial Rubor - week 48 (n=39,21): number analyzed (Participants) | 39 | 21
  Facial Rubor - week 48 (n=39,21) | 37 | 21
  Hirsutism - week 48 (n=33,15): number analyzed (Participants) | 33 | 15
  Hirsutism - week 48 (n=33,15) | 29 | 15
  Striae - week 48 (n=38,21): number analyzed (Participants) | 38 | 21
  Striae - week 48 (n=38,21) | 38 | 21
  Supraclavicular Fat Pad - week 48 (n=39,22): number analyzed (Participants) | 39 | 22
  Supraclavicular Fat Pad - week 48 (n=39,22) | 38 | 22
  Dorsal Fat Pad - week 48 (n=38,22): number analyzed (Participants) | 38 | 22
  Dorsal Fat Pad - week 48 (n=38,22) | 36 | 20
  Proximal Muscle Atrophy - week 48 (n=39,22): number analyzed (Participants) | 39 | 22
  Proximal Muscle Atrophy - week 48 (n=39,22) | 35 | 21
  Central Obesity - week 48 (n=39,22): number analyzed (Participants) | 39 | 22
  Central Obesity - week 48 (n=39,22) | 35 | 21
  Ecchymoses - week 48 (n=39,21): number analyzed (Participants) | 39 | 21
  Ecchymoses - week 48 (n=39,21) | 38 | 20

26. Secondary Outcome: Change From Baseline in Standardized Health Related Quality of Life Score, Using Cushing Disease-specific Quality of Life Patient Reported Outcome (PRO) Assessment
Description: The CushingQoL is a valid and reliable disease-specific QoL questionnaire which assesses health-related quality of life (HRQoL) in patients with Cushing's syndrome and has been validated in patients with Cushing's disease. The CushingQoL consists of questions reflecting dimensions of HRQoL related to physical aspects (e.g. 'I bruise easily'), psychological aspects (e.g. 'I am more irritable, I have sudden mood swings and angry outbursts'), and social aspects (e.g. 'I have had to give up my social or leisure activities due to my illness').
  The questionnaire consists of 12 items measured on a five point Likert-type scale assessing how often or how much each item has been related to the patient's Cushing's disease in the previous week. The raw score is calculated by summing the individual item scores prior to being standardized so that the total score ranges from 0 to 100. Increases from baseline are indicative of an improvement.
Time Frame: Baseline to Week 12 and 48, Week 12 to Week 36, Week 36 to Week 48.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
Scores on a scale
  Actual - Baseline (n=48,25) | 49.1 (19.60) | 56.9 (18.99)
  Actual Change from Baseline at Week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Actual Change from Baseline at Week 12 (n=46,24) | 6.2 (14.85) | 8.6 (12.06)
  Actual Change from Baseline at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Baseline at Week 48 (n=42,22) | 11.7 (16.30) | 12.8 (14.24)
  Actual Change from Week 12 at Week 36 (n=44,23): number analyzed (Participants) | 44 | 23
  Actual Change from Week 12 at Week 36 (n=44,23) | 4.7 (9.01) | -0.5 (9.99)
  Actual Change from Week 36 at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Week 36 at Week 48 (n=42,22) | 0.1 (8.43) | 2.5 (7.52)

27. Secondary Outcome: Change From Baseline in Standardized Psychosocial Issues Score, Using Cushing Disease-specific Quality of Life Patient Reported Outcome (PRO) Assessment
Description: as for outcome 26
Time Frame: Baseline to Week 12 and 48, Week 12 to Week 36, Week 36 to Week 48.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
Scores on a scale
  Actual - baseline (n=48,25) | 49.9 (20.34) | 56.7 (21.11)
  Actual Change from Baseline at Week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Actual Change from Baseline at Week 12 (n=46,24) | 6.1 (17.21) | 9.6 (13.61)
  Actual Change from Baseline at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Baseline at Week 48 (n=42,22) | 11.1 (17.84) | 13.0 (16.30)
  Actual Change from Week 12 at Week 36 (n=44,23): number analyzed (Participants) | 44 | 23
  Actual Change from Week 12 at Week 36 (n=44,23) | 4.1 (9.94) | -1.3 (12.36)
  Actual Change from Week 36 at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Week 36 at Week 48 (n=42,22) | 0.1 (9.60) | 2.4 (8.96)

28. Secondary Outcome: Change From Baseline in Standardized Physical Problems Score, Using Cushing Disease-specific Quality of Life Patient Reported Outcome (PRO) Assessment
Description: as for outcome 26
Time Frame: Baseline to Week 12 and 48, Week 12 to Week 36, Week 36 to Week 48.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
Scores on a scale
  Actual - baseline (n=48,25) | 46.9 (22.32) | 57.7 (21.91)
  Actual Change from Baseline at Week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Actual Change from Baseline at Week 12 (n=46,24) | 6.3 (13.29) | 5.6 (13.38)
  Actual Change from Baseline at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Baseline at Week 48 (n=42,22) | 13.3 (19.83) | 12.1 (15.59)
  Actual Change from Week 12 at Week 36 (n=44,23): number analyzed (Participants) | 44 | 23
  Actual Change from Week 12 at Week 36 (n=44,23) | 6.6 (12.40) | 2.2 (12.11)
  Actual Change from Week 36 at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Week 36 at Week 48 (n=42,22) | 23.59 (11.27) | 2.7 (12.17)

29. Secondary Outcome: Change From Baseline in EQ-5D-5L Utility Index
Description: EQ-5D-5L Utility Index:
  The EQ-5D-5L questionnaire is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L measures 5 items on mobility, self-care, usual activities, pain/discomfort, anxiety/depression, measured on 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. A utility index can be computed from the EQ 5D-5L descriptive system with utility scores ranging from -0.281 (worst imaginable health state) to 1 (best imaginable health state), with -0.281 representing an "unconscious" health state. A single index value is analyzed for the EQ-5D-5L score. An increase from baseline in the EQ-ED-5L utility index is indicative of an improvement.
Time Frame: Baseline to Week 12 and 48, Week 12 to Week 36, Week 36 to Week 48.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 24
Scores on a scale
  Actual - baseline (n=48,24) | 0.825 (0.1486) | 0.903 (0.1125)
  Actual Change from Baseline at Week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Actual Change from Baseline at Week 12 (n=46,24) | -0.000 (0.1402) | 0.021 (0.0771)
  Actual Change from Baseline at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Baseline at Week 48 (n=42,22) | 0.044 (0.1393) | 0.033 (0.0826)
  Actual Change from Week 12 at Week 36 (n=44,23): number analyzed (Participants) | 44 | 23
  Actual Change from Week 12 at Week 36 (n=44,23) | 0.025 (0.1283) | 0.010 (0.0487)
  Actual Change from Week 36 at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Week 36 at Week 48 (n=42,22) | 0.023 (0.0762) | -0.008 (0.0367)

30. Secondary Outcome: Change From Baseline in EQ-5D VAS
Description: The EQ-5D-5L also includes a 20 cm vertical, VAS (visual analogue scale) with a scale of 0-100, with endpoints labeled 100='the best health you can imagine' and 0='the worst health you can imagine'. A single index value is analyzed for the EQ-5D-5L VAS score. An increase from baseline in the EQ-ED-5L VAS is indicative of an improvement.
Time Frame: Baseline to Week 12 and 48, Week 12 to Week 36, Week 36 to Week 48.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 24
Scores on a scale
  Actual - baseline (n=48,23): number analyzed (Participants) | 48 | 23
  Actual - baseline (n=48,23) | 70.3 (17.26) | 76.7 (17.88)
  Actual Change from Baseline at week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Actual Change from Baseline at week 12 (n=46,24) | 0.5 (13.57) | -0.3 (10.52)
  Actual Change from Baseline at week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Baseline at week 48 (n=42,22) | 9.4 (13.13) | 5.8 (9.45)
  Actual Change from Week 12 at Week 36 (n=44,23): number analyzed (Participants) | 44 | 23
  Actual Change from Week 12 at Week 36 (n=44,23) | 6.0 (11.08) | 3.7 (9.29)
  Actual Change from Week 36 at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Week 36 at Week 48 (n=42,22) | 3.2 (8.40) | -0.8 (4.44)

31. Secondary Outcome: Change From Baseline in Beck Depression Inventory-II - Total Score Derived
Description: The Beck Depression Inventory II (BDI-II) is a patient reported instrument that consists of 21 items designed to assess the intensity of depression in clinical and normal patients in the preceding two weeks. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression. A global score ranges from 0 to 63 and is calculated with a higher score representing a greater level of depression. The following scoring guidelines for interpretation of BDI-II have been suggested (Smarr, 2011): Minimal range =0-13, Mild depression =14-19, Moderate depression =20-28 and Severe depression = 29-63. A reduction from baseline in BDI-II is indicative of an improvement.
Time Frame: Baseline to Week 12 and 48, Week 12 to Week 36, Week 36 to Week 48.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
Scores on a scale
  Actual - baseline (n=48,25) | 12.2 (10.22) | 8.4 (7.82)
  Actual Change from Baseline at Week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Actual Change from Baseline at Week 12 (n=46,24) | -1.4 (7.99) | -3.9 (5.42)
  Actual Change from Baseline at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Baseline at Week 48 (n=42,22) | -4.3 (7.52) | -4.0 (7.70)
  Actual Change from Week 12 at Week 36 (n=44,23): number analyzed (Participants) | 44 | 23
  Actual Change from Week 12 at Week 36 (n=44,23) | -2.0 (4.70) | 0.6 (6.29)
  Actual Change from Week 36 at Week 48 (n=42,22): number analyzed (Participants) | 42 | 22
  Actual Change from Week 36 at Week 48 (n=42,22) | -1.1 (4.83) | -0.4 (3.39)

32. Secondary Outcome: Change From Baseline in Serum Cortisol
Description: Change from baseline in serum cortisol
Time Frame: Baseline, Week 12, Week 36, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 47 | 25
nmol/L
  Baseline - actual (n=47,25) | 565.8 (169.01) | 486.1 (198.12)
  Actual Change from Baseline at Week 12 (n=44,24): number analyzed (Participants) | 44 | 24
  Actual Change from Baseline at Week 12 (n=44,24) | -276.0 (178.43) | 73.0 (185.29)
  Actual Change from Baseline at Week 36 (n=42,25): number analyzed (Participants) | 42 | 25
  Actual Change from Baseline at Week 36 (n=42,25) | -267.0 (174.18) | -157.8 (225.56)
  Actual Change from Baseline at Week 48 (n=41,22): number analyzed (Participants) | 41 | 22
  Actual Change from Baseline at Week 48 (n=41,22) | -210.7 (161.07) | -131.0 (236.88)

33. Secondary Outcome: Change From Baseline in Late Night Saliva Cortisol
Description: Change from baseline in late night saliva cortisol (nmol/L)
Time Frame: Baseline, Week 12, Week 36, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
nmol/L
  Baseline - actual (n=48,25) | 11.7 (28.68) | 9.0 (6.74)
  Actual Change from Baseline at Week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Actual Change from Baseline at Week 12 (n=46,24) | -8.5 (29.60) | 1.3 (8.87)
  Actual Change from Baseline at Week 36 (n=42,25): number analyzed (Participants) | 42 | 25
  Actual Change from Baseline at Week 36 (n=42,25) | -9.6 (30.82) | -5.8 (6.84)
  Actual Change from Baseline at Week 48 (n=41,22): number analyzed (Participants) | 41 | 22
  Actual Change from Baseline at Week 48 (n=41,22) | -9.3 (29.05) | -5.0 (5.75)

34. Secondary Outcome: Change From Baseline in Morning Saliva Cortisol
Description: Change from baseline in morning saliva cortisol (nmol/L)
Time Frame: Baseline, Week 12, Week 36, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 48 | 25
nmol/L
  Baseline - actual (n=48,25) | 17.2 (30.00) | 14.1 (12.29)
  Actual Change from Baseline at Week 12 (n=46,24): number analyzed (Participants) | 46 | 24
  Actual Change from Baseline at Week 12 (n=46,24) | -11.6 (30.05) | -0.3 (11.21)
  Actual Change from Baseline at Week 36 (n=40,25): number analyzed (Participants) | 40 | 25
  Actual Change from Baseline at Week 36 (n=40,25) | -11.8 (30.74) | -9.3 (11.82)
  Actual Change from Baseline at Week 48 (n=41,22): number analyzed (Participants) | 41 | 22
  Actual Change from Baseline at Week 48 (n=41,22) | -11.8 (31.74) | -6.0 (10.97)

35. Secondary Outcome: Change From Baseline in Hair Cortisol Levels
Description: Change from baseline in hair cortisol levels
Time Frame: Baseline, Week 26, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mg
Arm/Group | Osilodrostat Group | Osilodrostat Placebo Group
Number analyzed (Participants) | 19 | 9
pg/mg
  Baseline - actual (n=19,9) | 38.9 (37.48) | 10.5 (10.47)
  Actual Change from Baseline at Week 26 (n=16,7): number analyzed (Participants) | 16 | 7
  Actual Change from Baseline at Week 26 (n=16,7) | -15.8 (32.83) | -1.1 (12.72)
  Actual Change from Baseline at Week 48 (n=14,6): number analyzed (Participants) | 14 | 6
  Actual Change from Baseline at Week 48 (n=14,6) | -17.8 (26.66) | -9.7 (8.90)

36. Secondary Outcome: Plasma Osilodrostat Concentrations (ng/mL)
Description: Plasma osilodrostat concentrations (ng/mL)
Time Frame: pre-dose and 1-2hrs post dose at weeks 1, 2, 5, 8, 12, 14, 20, 26
Population: Pharmacokinetic Analysis Set (PAS): comprises all participants who received at least one dose of osilodrostat and have at least one evaluable pharmacokinetic concentration (post-first-dose) at any visit. The number analyzed varied from one visit to another because of missed visits, missed assessments, early discontinuation from the study, and completion of the extension phase. Note that participants took several different doses of study medication in this dose titration study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Osilodrostat Incident Dose 1mg: Participants received 1mg of osilodrostat.
- Osilodrostat Incident Dose 2mg: Participants received 2mg of osilodrostat.
- Osilodrostat Incident Dose 5mg: Participants received 5mg of osilodrostat.
Arm/Group | Osilodrostat Incident Dose 1mg | Osilodrostat Incident Dose 2mg | Osilodrostat Incident Dose 5mg
Number analyzed (Participants) | 16 | 55 | 29
ng/mL
  week 1 1-2 hrs post dose (n=1,43,0): number analyzed (Participants) | 1 | 43 | 0
  week 1 1-2 hrs post dose (n=1,43,0) | 3.85 (NA) — Geometric Coefficient of Variation is not applicable when 1 participant is analyzed | 7.29 (101.0) |
  week 2 0 hrs pre dose (n=0,41,0): number analyzed (Participants) | 0 | 41 | 0
  week 2 0 hrs pre dose (n=0,41,0) |  | 2.19 (107.5) |
  week 2 1-2 hrs post dose (n=0,42,0): number analyzed (Participants) | 0 | 42 | 0
  week 2 1-2 hrs post dose (n=0,42,0) |  | 9.76 (53.4) |
  week 5 pre dose (n=2,18,17): number analyzed (Participants) | 2 | 18 | 17
  week 5 pre dose (n=2,18,17) | 0.576 (141.9) | 2.07 (82.1) | 5.06 (109.6)
  week 5 1-2 hrs post dose (n=2,9,29): number analyzed (Participants) | 2 | 9 | 29
  week 5 1-2 hrs post dose (n=2,9,29) | 3.64 (60.5) | 11.1 (31.5) | 25.8 (84.4)
  week 8 0 hrs pre dose (n=2,4,13): number analyzed (Participants) | 2 | 4 | 13
  week 8 0 hrs pre dose (n=2,4,13) | 0.971 (76.7) | 2.64 (53.7) | 4.99 (55.6)
  week 8 1-2 hrs post dose (n=3,6,14): number analyzed (Participants) | 3 | 6 | 14
  week 8 1-2 hrs post dose (n=3,6,14) | 3.70 (47.6) | 8.31 (45.6) | 23.3 (68.1)
  week 12 0 hrs pre dose (n=2,8,11): number analyzed (Participants) | 2 | 8 | 11
  week 12 0 hrs pre dose (n=2,8,11) | 1.55 (3.7) | 2.45 (39.2) | 5.03 (74.6)
  week 12 1-2 hrs post dose (n=4,34,0): number analyzed (Participants) | 4 | 34 | 0
  week 12 1-2 hrs post dose (n=4,34,0) | 4.93 (32.0) | 11.7 (78.9) |
  week 14 0 hrs pre dose (n=4,55,0): number analyzed (Participants) | 4 | 55 | 0
  week 14 0 hrs pre dose (n=4,55,0) | 0.974 (129.7) | 1.96 (74.9) |
  week 14 1-2 hrs post dose (n=6,49,6): number analyzed (Participants) | 6 | 49 | 6
  week 14 1-2 hrs post dose (n=6,49,6) | 3.74 (161.4) | 9.69 (35.8) | 22.6 (37.8)
  week 20 0 hrs pre dose (n=10,19,15): number analyzed (Participants) | 10 | 19 | 15
  week 20 0 hrs pre dose (n=10,19,15) | 1.63 (71.1) | 1.95 (68.1) | 6.21 (74.3)
  week 20 1-2 hrs post dose (n=13,18,12): number analyzed (Participants) | 13 | 18 | 12
  week 20 1-2 hrs post dose (n=13,18,12) | 6.09 (27.3) | 8.66 (94.0) | 26.0 (99.3)
  week 26 0 hrs pre dose (n=12,13,10): number analyzed (Participants) | 12 | 13 | 10
  week 26 0 hrs pre dose (n=12,13,10) | 1.77 (86.4) | 2.12 (77.8) | 6.89 (85.1)
  week 26 1-2 hrs post dose (n=16,14,10): number analyzed (Participants) | 16 | 14 | 10
  week 26 1-2 hrs post dose (n=16,14,10) | 5.28 (31.5) | 8.04 (50.7) | 33.1 (31.4)

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 8 weeks post treatment, up to maximum duration of 116.7 weeks.
Groups:
- Placebo Controlled Period - Osilodrostat Arm.: All data while on osilodrostat treatment up to week 12 in participants initially randomized to osilodrostat.
- Placebo Controlled Period - Placebo Arm.: All data while on placebo treatment up to week 12 in participants initially randomized to placebo.
- Overall Study Period - Osilodrostat Arm.: All data while on osilodrostat treatment from randomization up to end-of-study in participants initially randomized to osilodrostat.
- Overall Study Period - Placebo Arm.: All data while on osilodrostat treatment from Week 12 up to end-of-study in participants initially randomized to placebo.
- Overall Study Period - All Participants.: All data while on osilodrostat treatment up to end-of-study in all randomized participants, excluding data while on placebo from participants initially randomized to placebo.
Arm/Group | Placebo Controlled Period - Osilodrostat Arm. | Placebo Controlled Period - Placebo Arm. | Overall Study Period - Osilodrostat Arm. | Overall Study Period - Placebo Arm. | Overall Study Period - All Participants.
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/25 | 0/48 | 0/25 | 0/73
Serious Adverse Events (participants affected / at risk) | 2/48 | 1/25 | 10/48 | 0/25 | 10/73
Other Adverse Events (participants affected / at risk) | 45/48 | 21/25 | 47/48 | 24/25 | 71/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Controlled Period - Osilodrostat Arm. (N=48) | Placebo Controlled Period - Placebo Arm. (N=25) | Overall Study Period - Osilodrostat Arm. (N=48) | Overall Study Period - Placebo Arm. (N=25) | Overall Study Period - All Participants. (N=73)
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 3 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Conjunctival laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Retinal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 1 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Cerebral vascular occlusion (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Controlled Period - Osilodrostat Arm. (N=48) | Placebo Controlled Period - Placebo Arm. (N=25) | Overall Study Period - Osilodrostat Arm. (N=48) | Overall Study Period - Placebo Arm. (N=25) | Overall Study Period - All Participants. (N=73)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 1 | 3
Palpitations (Cardiac disorders) | 0 | 2 | 2 | 0 | 2
Tachycardia (Cardiac disorders) | 6 | 0 | 8 | 1 | 9
Adrenal insufficiency (Endocrine disorders) | 7 | 0 | 12 | 6 | 18
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 4 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 10 | 2 | 12
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 10 | 0 | 14 | 3 | 17
Nausea (Gastrointestinal disorders) | 15 | 3 | 22 | 5 | 27
Vomiting (Gastrointestinal disorders) | 5 | 0 | 9 | 0 | 9
Asthenia (General disorders) | 11 | 0 | 15 | 2 | 17
Fatigue (General disorders) | 12 | 4 | 23 | 6 | 29
Oedema peripheral (General disorders) | 5 | 0 | 12 | 0 | 12
Pyrexia (General disorders) | 2 | 0 | 5 | 0 | 5
Gastroenteritis (Infections and infestations) | 1 | 0 | 4 | 0 | 4
Influenza (Infections and infestations) | 2 | 0 | 4 | 0 | 4
Laryngitis (Infections and infestations) | 0 | 0 | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 2 | 4
Oral herpes (Infections and infestations) | 1 | 0 | 3 | 0 | 3
Pharyngitis (Infections and infestations) | 1 | 0 | 5 | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 0 | 12 | 4 | 16
Urinary tract infection (Infections and infestations) | 4 | 0 | 8 | 4 | 12
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 4 | 0 | 4
Alanine aminotransferase increased (Investigations) | 2 | 2 | 3 | 3 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 3 | 5
Blood cholesterol increased (Investigations) | 2 | 1 | 3 | 0 | 3
Blood potassium decreased (Investigations) | 1 | 1 | 2 | 2 | 4
Blood pressure increased (Investigations) | 1 | 1 | 3 | 0 | 3
Blood testosterone increased (Investigations) | 5 | 0 | 13 | 5 | 18
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 2 | 2
Renin increased (Investigations) | 1 | 0 | 1 | 4 | 5
Weight decreased (Investigations) | 2 | 0 | 3 | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 18 | 4 | 24 | 10 | 34
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 1 | 6 | 0 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 6 | 2 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 3 | 26 | 7 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 8 | 2 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 1 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 1 | 15 | 3 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 2 | 5
Dizziness (Nervous system disorders) | 9 | 4 | 19 | 3 | 22
Headache (Nervous system disorders) | 7 | 6 | 17 | 8 | 25
Paraesthesia (Nervous system disorders) | 0 | 0 | 4 | 0 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 2 | 4
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 9 | 1 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 1 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 1 | 4
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 4
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 6 | 1 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 0 | 7 | 2 | 9
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 1 | 4
Hypertension (Vascular disorders) | 7 | 7 | 12 | 4 | 16
Hypotension (Vascular disorders) | 5 | 0 | 9 | 3 | 12
Orthostatic hypotension (Vascular disorders) | 4 | 0 | 7 | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT02697734/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT02697734/SAP_001.pdf